CLINICAL TRIAL: NCT03037632
Title: Precision Medicine for Dilated Cardiomyopathy in European and African Ancestry
Brief Title: DCM Precision Medicine Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ray Hershberger (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor-Investigator, Ray Hershberger, MD, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015H0309; R01HL128857 (NIH)
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinded until intervention is assigned to subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Communication Tool (Experimental)
  Interventions: Behavioral: Family Heart Talk Booklet
- No Communication Tool (No Intervention)

INTERVENTIONS:
Behavioral: Family Heart Talk Booklet
  Arms: Communication Tool

SUMMARY:
The aims of the DCM Precision Medicine Study are to test the hypothesis that DCM has substantial genetic basis and to evaluate the effectiveness of a family communication intervention in improving the uptake and impact of family member clinical screening.

DETAILED DESCRIPTION:
Dilated cardiomyopathy of unknown cause (DCM), known clinically as idiopathic dilated cardiomypathy, is the most common cardiomyopathy and is the leading cause of heart transplantation. DCM affects approximately one million individuals, and so has a major impact on US public health. DCM is commonly asymptomatic until very late in its course when it causes heart failure, disability, and death. Because of its clinical course, any means to identify patients at risk for DCM or to detect DCM in its asymptomatic phase could provide enormous opportunity for intervention to extend lives and prevent late-stage disease. Within this paradigm precision medicine for DCM could greatly impact health care outcomes and costs. Recent advances in DCM genetics have introduced these possibilities, but unresolved questions of familial recurrence risk, genetic etiology, racial differences, and family-based screening must be addressed to move ahead. The central hypothesis of this study, based on published studies of the investigative group, states that DCM has substantial genetic basis. For this study the investigators hypothesize that: (a) 35% of probands of both European and African ancestry (EA/AA) will be classified as familial in a cohort recruited in a multicenter US consortium and given explicit recommendations and assistance to achieve the clinical screening of relatives; (b) approximately 40% of DCM probands, whether categorized as familial or non-familial, or as EA or AA, will have pathogenic or likely pathogenic variants in genes previously implicated in DCM; and (c) a tailored intervention to help DCM probands communicate DCM risk to their family members will improve the uptake and impact of necessary clinical and genetic testing. To test these hypotheses, the investigators propose to: (1) estimate and compare the frequencies of EA and AA DCM probands classified as having familial DCM; (2) estimate and compare the proportions of probands with an identifiable genetic cause of DCM in groups defined by proband classification (familial/non-familial) and ancestry (EA/AA); and (3) evaluate the impact of a randomized intervention to aid and direct family communication on participation of at-risk family members in clinical screening and appropriate follow-up surveillance for DCM. These aims will be accomplished by recruiting a cohort of 1300 DCM probands (600 EA, 600 AA, 100 Hispanic ethnicity), performing cardiovascular clinical screening of 2600 family members, performing genetic testing of probands and affected family members by exome sequencing, returning genetic results, and randomizing probands to an intervention to improve family communication regarding DCM risk. Proving these hypotheses would be transformative for the field: rather than viewing DCM as only a clinical diagnosis, cardiovascular professionals would understand DCM as a genetic disease that should be managed using genetic diagnostic and family-based preventive strategies. These study results would make precision medicine for DCM a reality.

ELIGIBILITY:
Inclusion Criteria:

* Meeting criteria for dilated cardiomyopathy (DCM) :

  * Left ventricular ejection fraction <50%
  * Left ventricular enlargement (A left ventricular end-diastolic dimension > 95%tile population standard based on gender and height).
* Detectable causes of cardiomyopathy, except genetic, excluded beyond a reasonable doubt at the time of DCM diagnosis (that is, meeting clinical criteria for idiopathic DCM)
* Any age (including children)
* Non-Hispanic and Hispanic ethnicity
* All races (PI pre-approval required for recruitment beyond pre-specified recruitment targets).
* Ability to give informed consent
* Ability to communicate in English (except Spanish language at sites approved to recruit individuals of Hispanic ethnicity)
* Willingness to participate in a family-based study (patient willing to work with a clinical site and/or OSU to facilitate the recruitment and enrollment of family members to the study).

Exclusion Criteria:

* Coronary artery disease (CAD) causing ischemic cardiomyopathy (> 50% narrowing, any major epicardial coronary artery)
* Primary valvular disease
* Adriamycin or other cardiotoxic drug exposure
* Other forms of cardiomyopathy: Hypertrophic, Restrictive, or Arrhythmogenic Right Ventricular Dysplasia/Cardiomyopathy
* Congenital heart disease
* Other detectable causes of dilated cardiomyopathy, including sarcoid and hemochromatosis.
* Other active multi-system disease that may cause DCM (e.g., active connective tissue disease).
* Severe and untreated or untreatable hypertension (systolic blood pressures routinely greater than 180 mm Hg and/or diastolic blood pressures greater than 120 mm Hg, and if resistant to multidrug treatment).
* However, conventional risk factors for DCM, including obesity, routinely treated hypertension, alcohol use, pregnancy or the peri-partum period, or left ventricular noncompaction, will NOT be considered exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6500 (Estimated)
Dates: Start 2016-06-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Family clinical screening completed within 12 months from proband enrollment. | 12 months from proband enrollment.
  The probability that a living first-degree relative (FDR) without a previous definitive DCM diagnosis completes clinical screening for DCM within 12 months after proband recruitment
Living first-degree relative adheres to cardiovascular surveillance recommendations after return of genetic results. | 2.5 years
  The probability that a living first-degree relative adheres to surveillance recommendations within 15 months after the proband receives individual genetic test information.

CONTACTS AND LOCATIONS:
Overall Officials: Ray Hershberger, MD, Principal Investigator — Ohio State University
Locations (26):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Medstar Washington Hospital Center (DC), Washington D.C., District of Columbia
  - South Miami Heart Center, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Louisiana State University Health Sciences Center in New Orleans, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Heart and Vascular Institute, Fairfax, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cowan JR, Hershberger RE. Transcriptomics and Beyond in Dilated Cardiomyopathy. JACC Basic Transl Sci. 2023 Apr 24;8(4):419-421. doi: 10.1016/j.jacbts.2023.01.016. eCollection 2023 Apr. PMID 37138804
- [Background] Jordan E, Ni H, Parker P, Kinnamon DD, Owens A, Lowes B, Shenoy C, Martin CM, Judge DP, Fishbein DP, Stoller D, Minami E, Kransdorf E, Smart F, Haas GJ, Huggins GS, Ewald GA, Diamond J, Wilcox JE, Jimenez J, Wang J, Tallaj J, Drazner MH, Hofmeyer M, Wheeler MT, Pinzon OW, Shah P, Gottlieb SS, Katz S, Shore S, Tang WHW, Hershberger RE; DCM Precision Medicine study of the DCM Consortium. Implementing Precision Medicine for Dilated Cardiomyopathy: Insights from The DCM Consortium. medRxiv [Preprint]. 2024 Nov 26:2024.11.22.24317816. doi: 10.1101/2024.11.22.24317816. PMID 39649582
- [Background] Kransdorf EP, Jain R, Mead JO, Haas G, Hofmeyer M, Ewald GA, Diamond J, Owens A, Lowes B, Stoller D, Tang WHW, Drazner MH, Martin CM, Shah P, Tallaj J, Katz S, Jimenez J, Shore S, Smart F, Wang J, Gottlieb SS, Judge DP, Huggins GS, Cowan J, Parker P, Cao J, Hurst NS, Jordan E, Ni H, Kinnamon DD, Hershberger RE. Evaluation of Women with Peripartum or Dilated Cardiomyopathy and Their First-Degree Relatives: The DCM Precision Medicine Study. medRxiv [Preprint]. 2025 Jun 8:2025.02.18.25322501. doi: 10.1101/2025.02.18.25322501. PMID 40034776
- [Background] Hershberger RE, Ni H. Systemic Immune-Mediated Diseases and Dilated Cardiomyopathy. JACC Heart Fail. 2025 Jan;13(1):146-148. doi: 10.1016/j.jchf.2024.11.002. No abstract available. PMID 39779179
- [Background] Ni H, Jordan E, Cao J, Kinnamon DD, Gottlieb SS, Hofmeyer M, Jimenez J, Judge DP, Kransdorf E, Morris AA, Owens A, Shah P, Tang WHW, Wang J, Hershberger RE. Knowledge of Genome Sequencing and Trust in Medical Researchers Among Patients of Different Racial and Ethnic Groups With Idiopathic Dilated Cardiomyopathy. JAMA Cardiol. 2023 Jan 1;8(1):33-42. doi: 10.1001/jamacardio.2022.4132. PMID 36383367
- [Background] Jordan ES, Grover PL, Lin J, Starkey CA, Finley EA, Ni H, Hershberger RE. The DCM Project Portal: A direct-to-participant platform of The DCM Research Project. Am Heart J Plus. 2024 Feb;38:100356. doi: 10.1016/j.ahjo.2023.100356. Epub 2023 Dec 27. PMID 38348286
- [Background] Hofmeyer M, Haas GJ, Jordan E, Cao J, Kransdorf E, Ewald GA, Morris AA, Owens A, Lowes B, Stoller D, Wilson Tang WH, Garg S, Trachtenberg BH, Shah P, Pamboukian SV, Sweitzer NK, Wheeler MT, Wilcox JE, Katz S, Pan S, Jimenez J, Smart F, Wang J, Gottlieb SS, Judge DP, Moore CK, Huggins GS, Kinnamon DD, Ni H, Hershberger RE; DCM Precision Medicine Study of the DCM Consortium. Rare Variant Genetics and Dilated Cardiomyopathy Severity: The DCM Precision Medicine Study. Circulation. 2023 Sep 12;148(11):872-881. doi: 10.1161/CIRCULATIONAHA.123.064847. Epub 2023 Aug 29. PMID 37641966
- [Background] Kinnamon DD, Morales A, Bowen DJ, Burke W, Hershberger RE; DCM Consortium*. Toward Genetics-Driven Early Intervention in Dilated Cardiomyopathy: Design and Implementation of the DCM Precision Medicine Study. Circ Cardiovasc Genet. 2017 Dec;10(6):e001826. doi: 10.1161/CIRCGENETICS.117.001826. PMID 29237686
- [Background] Morales A, Kinnamon DD, Jordan E, Platt J, Vatta M, Dorschner MO, Starkey CA, Mead JO, Ai T, Burke W, Gastier-Foster J, Jarvik GP, Rehm HL, Nickerson DA, Hershberger RE; DCM Precision Medicine study of the DCM Consortium; DCM Consortium institutions and personnel participating in this study: Study Principal Investigator and Co-Investigators,DCM Consortium Clinical Site Principal Investigators and Clinical Site Other Significant Contributors (OSC). The following clinical sites and individuals contributed to the submission of RO 1 H L 128857 as Site Principal Investigators (Site Pl) or as Other Significant Contributors (OSC),Dr. Huggins also served as study co-principal investigator,The following clinical site was added following approval of NHGRI supplemental funding but prior to initiation of enrollment,The following clinical sites were added following study activation. Variant Interpretation for Dilated Cardiomyopathy: Refinement of the American College of Medical Genetics and Genomics/ClinGen Guidelines for the DCM Precision Medicine Study. Circ Genom Precis Med. 2020 Apr;13(2):e002480. doi: 10.1161/CIRCGEN.119.002480. Epub 2020 Mar 11. PMID 32160020
- [Background] Kinnamon DD, Jordan E, Haas GJ, Hofmeyer M, Kransdorf E, Ewald GA, Morris AA, Owens A, Lowes B, Stoller D, Tang WHW, Garg S, Trachtenberg BH, Shah P, Pamboukian SV, Sweitzer NK, Wheeler MT, Wilcox JE, Katz S, Pan S, Jimenez J, Aaronson KD, Fishbein DP, Smart F, Wang J, Gottlieb SS, Judge DP, Moore CK, Mead JO, Huggins GS, Ni H, Burke W, Hershberger RE; DCM Precision Medicine Study of the DCM Consortium. Effectiveness of the Family Heart Talk Communication Tool in Improving Family Member Screening for Dilated Cardiomyopathy: Results of a Randomized Trial. Circulation. 2023 Apr 25;147(17):1281-1290. doi: 10.1161/CIRCULATIONAHA.122.062507. Epub 2023 Mar 20. PMID 36938756
- [Background] Haas GJ, Zareba KM, Ni H, Bello-Pardo E, Huggins GS, Hershberger RE; Study Principal Investigator (PI) and Co-Investigators: The Ohio State University. Validating an Idiopathic Dilated Cardiomyopathy Diagnosis Using Cardiovascular Magnetic Resonance: The Dilated Cardiomyopathy Precision Medicine Study. Circ Heart Fail. 2022 May;15(5):e008877. doi: 10.1161/CIRCHEARTFAILURE.121.008877. Epub 2022 Mar 4. PMID 35240856
- [Background] Huggins GS, Kinnamon DD, Haas GJ, Jordan E, Hofmeyer M, Kransdorf E, Ewald GA, Morris AA, Owens A, Lowes B, Stoller D, Tang WHW, Garg S, Trachtenberg BH, Shah P, Pamboukian SV, Sweitzer NK, Wheeler MT, Wilcox JE, Katz S, Pan S, Jimenez J, Aaronson KD, Fishbein DP, Smart F, Wang J, Gottlieb SS, Judge DP, Moore CK, Mead JO, Ni H, Burke W, Hershberger RE; DCM Precision Medicine Study of the DCM Consortium. Prevalence and Cumulative Risk of Familial Idiopathic Dilated Cardiomyopathy. JAMA. 2022 Feb 1;327(5):454-463. doi: 10.1001/jama.2021.24674. PMID 35103767
- [Background] Burke W, Hovick SR, Jordan E, Ni H, Kinnamon DD, Hershberger RE. Communal Coping as a Strategy to Enhance Family Engagement in Dilated Cardiomyopathy. Circ Genom Precis Med. 2022 Jun;15(3):e003541. doi: 10.1161/CIRCGEN.121.003541. Epub 2022 May 10. PMID 35536229
- [Background] Trachtenberg BH, Jimenez J, Morris AA, Kransdorf E, Owens A, Fishbein DP, Jordan E, Kinnamon DD, Mead JO, Huggins GS, Hershberger RE; DCM Precision Medicine Study of the DCM Consortium. TTR variants in patients with dilated cardiomyopathy: An investigation of the DCM Precision Medicine Study. Genet Med. 2022 Jul;24(7):1495-1502. doi: 10.1016/j.gim.2022.03.011. Epub 2022 Apr 18. PMID 35438637
- [Background] Hershberger RE, Cowan J, Jordan E, Kinnamon DD. The Complex and Diverse Genetic Architecture of Dilated Cardiomyopathy. Circ Res. 2021 May 14;128(10):1514-1532. doi: 10.1161/CIRCRESAHA.121.318157. Epub 2021 May 13. PMID 33983834
- [Background] Hershberger RE. The Evolving Science of Dilated Cardiomyopathy. J Am Coll Cardiol. 2021 Oct 26;78(17):1700-1702. doi: 10.1016/j.jacc.2021.08.038. No abstract available. PMID 34674814
- [Background] Ni H, Jordan E, Kinnamon DD, Cao J, Haas GJ, Hofmeyer M, Kransdorf E, Ewald GA, Morris AA, Owens A, Lowes B, Stoller D, Tang WHW, Garg S, Trachtenberg BH, Shah P, Pamboukian SV, Sweitzer NK, Wheeler MT, Wilcox JE, Katz S, Pan S, Jimenez J, Fishbein DP, Smart F, Wang J, Gottlieb SS, Judge DP, Moore CK, Huggins GS, Hershberger RE; DCM Precision Medicine Study of the DCM Consortium. Screening for Dilated Cardiomyopathy in At-Risk First-Degree Relatives. J Am Coll Cardiol. 2023 May 30;81(21):2059-2071. doi: 10.1016/j.jacc.2023.03.419. PMID 37225358
- [Background] Jordan E, Kinnamon DD, Haas GJ, Hofmeyer M, Kransdorf E, Ewald GA, Morris AA, Owens A, Lowes B, Stoller D, Tang WHW, Garg S, Trachtenberg BH, Shah P, Pamboukian SV, Sweitzer NK, Wheeler MT, Wilcox JE, Katz S, Pan S, Jimenez J, Fishbein DP, Smart F, Wang J, Gottlieb SS, Judge DP, Moore CK, Mead JO, Hurst N, Cao J, Huggins GS, Cowan J, Ni H, Rehm HL, Jarvik GP, Vatta M, Burke W, Hershberger RE; DCM Precision Medicine Study of the DCM Consortium. Genetic Architecture of Dilated Cardiomyopathy in Individuals of African and European Ancestry. JAMA. 2023 Aug 1;330(5):432-441. doi: 10.1001/jama.2023.11970. PMID 37526719
- [Derived] Ni H, Cao J, Kinnamon DD, Jordan E, Haas GJ, Hofmeyer M, Kransdorf EP, Diamond J, Owens A, Lowes B, Stoller D, Tang WHW, Drazner MH, Shah P, Wilcox JE, Katz SD, Jimenez J, Shore S, Judge DP, Mead JO, Cowan J, Parker PK, Huggins GS, Hershberger RE. Antecedent Flu-Like Illness and Onset of Idiopathic Dilated Cardiomyopathy: The DCM Precision Medicine Study. Circ Heart Fail. 2025 May;18(5):e012602. doi: 10.1161/CIRCHEARTFAILURE.124.012602. Epub 2025 Apr 14. PMID 40392911
- [Derived] Jimenez J, Ni H, Katz SD, Haas GJ, Cao J, Rubens M, Chaparro S, Saxena A, Hofmeyer M, Kransdorf E, Ewald GA, Morris AA, Owens A, Lowes B, Stoller D, Tang WHW, Shah P, Wilcox JE, Smart F, Wang J, Gottlieb SS, Judge DP, Mead JO, Hurst N, Parker PK, Huggins GS, Jordan E, Kinnamon DD, Hershberger RE; DCM Precision Medicine Study of the DCM Consortium. Alcohol Exposure Among Patients With Dilated Cardiomyopathy and Their First-Degree Relatives: The DCM Precision Medicine Study. Circ Genom Precis Med. 2025 Apr;18(2):e004946. doi: 10.1161/CIRCGEN.124.004946. Epub 2025 Mar 28. PMID 40151927
- [Derived] Wilcox JE, Beussink-Nelson L, Cao J, Kumar R, Jordan E, Ni H, Shah SJ, Hershberger RE, Kinnamon DD. Differences in Cardiac Mechanics among Genetically At-Risk First-Degree Relatives: The DCM Precision Medicine Study. medRxiv [Preprint]. 2023 Jun 4:2023.05.30.23290123. doi: 10.1101/2023.05.30.23290123. PMID 37398079
- See also: Additional information regarding DCM Precision Medicine Study information provided on website. — http://DCMProject.com